CLINICAL TRIAL: NCT05056077
Title: Optimizing Intervention Tools to Improve Nutrition and Physical Activity for Cancer Survivors (Tools To Be Fit)
Brief Title: Improving Nutrition and Physical Activity for Cancer Survivors (Tools To Be Fit)
Acronym: TTBF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of California, Davis (Other); Robert H. Lurie Cancer Center (Other); Dana-Farber Cancer Institute (Other); American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 21456; NCI-2021-09059 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R37CA248774 (NIH)
Record Dates: First submitted 2021-09-14; First posted 2021-09-24 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Bladder Cancer; Breast Cancer; Colon Cancer; Endometrial Cancer; Ovarian Cancer; Rectal Cancer; Prostate Cancer; Renal Cell Carcinoma; Kidney Cancer
Keywords: Cancer Survivors; Nutrition
MeSH Terms: conditions — Urinary Bladder Neoplasms; Breast Neoplasms; Colonic Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms; Rectal Neoplasms; Prostatic Neoplasms; Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Counseling; Early Intervention, Educational; Educational Status; Methods; Health Promotion; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (16):
- Condition I (text, health kit, health coach, support coach) (Experimental): Patients receive a personal report comparing their nutrition and physical activity to ACS guidelines and a booklet on nutrition and physical activity for patients with a history of cancer. Patients receive text messages and use digital health tool kit for 48 weeks. Patients also receive 13 health coaching sessions over 30-45 minutes each for 48 weeks. Support persons receive four coaching sessions lasting 30 minutes each, approximately every 12 weeks for 48 weeks.
  Interventions: Other: Counseling; Other: Educational Intervention; Behavioral: Health Education; Other: Health Promotion and Education - Direct Text Messaging; Other: Health Promotion and Education - Digital health tool kit; Other: Questionnaires
- Condition II (text, health kit, health coach) (Experimental): Patients receive a personal report comparing their nutrition and physical activity to ACS guidelines and a booklet on nutrition and physical activity for patients with a history of cancer cancer. Patients receive text messages and use digital health tool kit for 48 weeks. Patients also receive 13 health coaching sessions over 30 minutes each for 48 weeks.
  Interventions: Other: Educational Intervention; Behavioral: Health Education; Other: Health Promotion and Education - Direct Text Messaging; Other: Health Promotion and Education - Digital health tool kit; Other: Questionnaires
- Condition III (text, health kit, support coach) (Experimental): Patients receive a personal report comparing their nutrition and physical activity to ACS guidelines and a booklet on nutrition and physical activity for patients with a history of cancer. Patients receive text messages and use digital health tool kit for 48 weeks. Support persons receive four coaching sessions lasting 30 minutes each, approximately every 12 weeks for 48 weeks.
  Interventions: Other: Counseling; Other: Educational Intervention; Other: Health Promotion and Education - Direct Text Messaging; Other: Health Promotion and Education - Digital health tool kit; Other: Questionnaires
- Condition IV (text, health kit) (Experimental): Patients receive a personal report comparing their nutrition and physical activity to ACS guidelines and a booklet on nutrition and physical activity for patients with a history of cancer. Patients receive text messages and use digital health tool kit for 48 weeks.
  Interventions: Other: Educational Intervention; Other: Health Promotion and Education - Direct Text Messaging; Other: Health Promotion and Education - Digital health tool kit; Other: Questionnaires
- Condition IX (health kit, health coach, support coach) (Experimental): Patients receive a personal report comparing their nutrition and physical activity to ACS guidelines and a booklet on nutrition and physical activity for patients with a history of cancer. Patients use digital health tool kit for 48 weeks. Patients also receive 13 health coaching sessions over 30 minutes each for 48 weeks. Support persons receive four coaching sessions lasting 30 minutes each, approximately every 12 weeks for 48 weeks.
  Interventions: Other: Counseling; Other: Educational Intervention; Behavioral: Health Education; Other: Health Promotion and Education - Digital health tool kit; Other: Questionnaires
- Condition V (text, health coach, support coach) (Experimental): Patients receive a personal report comparing their nutrition and physical activity to ACS guidelines and a booklet on nutrition and physical activity for patients with a history of cancer. Patients receive text messages for 48 weeks. Patients also receive 15 health coaching sessions over 30 minutes each for 48 weeks. Support persons receive four coaching sessions lasting 30 minutes each, approximately every 12 weeks for 48 weeks.
  Interventions: Other: Counseling; Other: Educational Intervention; Behavioral: Health Education; Other: Health Promotion and Education - Direct Text Messaging; Other: Questionnaires
- Condition VI (text, health coach) (Experimental): Patients receive a personal report comparing their nutrition and physical activity to ACS guidelines and a booklet on nutrition and physical activity for patients with a history of cancer. Patients receive text messages for 48 weeks. Patients also receive 13 health coaching sessions over 30 minutes each for 48 weeks.
  Interventions: Other: Educational Intervention; Behavioral: Health Education; Other: Health Promotion and Education - Direct Text Messaging; Other: Questionnaires
- Condition VII (text, support coach) (Experimental): Patients receive a personal report comparing their nutrition and physical activity to ACS guidelines and a booklet on nutrition and physical activity for patients with a history of cancer. Patients receive text messages for 48 weeks. Support persons receive four coaching sessions lasting 30 minutes each, approximately every 12 weeks for 48 weeks.
  Interventions: Other: Counseling; Other: Educational Intervention; Other: Health Promotion and Education - Direct Text Messaging; Other: Questionnaires
- Condition VIII (text) (Experimental): Patients receive a personal report comparing their nutrition and physical activity to ACS guidelines and a booklet on nutrition and physical activity for patients with a history of cancer. Patients receive text messages for 48 weeks.
  Interventions: Other: Educational Intervention; Other: Health Promotion and Education - Direct Text Messaging; Other: Questionnaires
- Condition X (health kit, health coach) (Experimental): Patients receive a personal report comparing their nutrition and physical activity to ACS guidelines and a booklet on nutrition and physical activity for patients with a history of cancer. Patients use digital health tool kit for 48 weeks. Patients also receive 13 health coaching sessions over 30 minutes each for 48 weeks.
  Interventions: Other: Educational Intervention; Behavioral: Health Education; Other: Health Promotion and Education - Digital health tool kit; Other: Questionnaires
- Condition XI (health kit, support coach) (Experimental): Patients receive a personal report comparing their nutrition and physical activity to ACS guidelines and a booklet on nutrition and physical activity for patients with a history of cancer. Patients use digital health tool kit for 48 weeks. Support persons receive four coaching sessions lasting 30 minutes each, approximately every 12 weeks for 48 weeks.
  Interventions: Other: Counseling; Other: Educational Intervention; Other: Health Promotion and Education - Digital health tool kit; Other: Questionnaires
- Condition XII (health kit) (Experimental): Patients receive a personal report comparing their nutrition and physical activity to ACS guidelines and a booklet on nutrition and physical activity for patients with a history of cancer. Patients use digital health tool kit for 48 weeks.
  Interventions: Other: Educational Intervention; Other: Health Promotion and Education - Digital health tool kit; Other: Questionnaires
- Condition XIII (health coach, support coach) (Experimental): Patients receive a personal report comparing their nutrition and physical activity to ACS guidelines and a booklet on nutrition and physical activity for patients with a history of cancer. Patients receive 13 health coaching sessions over 30 minutes each for 48 weeks. Support persons receive four coaching sessions lasting 30 minutes each, approximately every 12 weeks for 48 weeks.
  Interventions: Other: Counseling; Other: Educational Intervention; Behavioral: Health Education; Other: Questionnaires
- Condition XIV (health coach) (Experimental): Patients receive a personal report comparing their nutrition and physical activity to ACS guidelines and a booklet on nutrition and physical activity for patients with a history of cancer. Patients receive 13 health coaching sessions over 30 minutes each for 48 weeks.
  Interventions: Other: Educational Intervention; Behavioral: Health Education; Other: Questionnaires
- Condition XV (support coach) (Experimental): Patients receive a personal report comparing their nutrition and physical activity to ACS guidelines and a booklet on nutrition and physical activity for patients with a history of cancer. Support persons receive four coaching sessions lasting 30 minutes each, approximately every 12 weeks for 48 weeks.
  Interventions: Other: Counseling; Other: Educational Intervention; Other: Questionnaires
- Condition XVI (study booklet) (Experimental): Patients receive a personal report comparing their nutrition and physical activity to ACS guidelines and a booklet on nutrition and physical activity for patients with a history of cancer.
  Interventions: Other: Educational Intervention; Other: Questionnaires

INTERVENTIONS:
Other: Counseling — Receive support person coaching
  Other Names: Counseling Intervention
  Arms: Condition I (text, health kit, health coach, support coach); Condition III (text, health kit, support coach); Condition IX (health kit, health coach, support coach); Condition V (text, health coach, support coach); Condition VII (text, support coach); Condition XI (health kit, support coach); Condition XIII (health coach, support coach); Condition XV (support coach)
Other: Educational Intervention — Receive personal report and booklet on nutrition and physical activity for patients with a history of cancer
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Behavioral: Health Education — Receive health coaching
  Other Names: Health Coaching
  Arms: Condition I (text, health kit, health coach, support coach); Condition II (text, health kit, health coach); Condition IX (health kit, health coach, support coach); Condition V (text, health coach, support coach); Condition VI (text, health coach); Condition X (health kit, health coach); Condition XIII (health coach, support coach); Condition XIV (health coach)
Other: Health Promotion and Education - Direct Text Messaging — Receive text messages
  Other Names: Text Messaging
  Arms: Condition I (text, health kit, health coach, support coach); Condition II (text, health kit, health coach); Condition III (text, health kit, support coach); Condition IV (text, health kit); Condition V (text, health coach, support coach); Condition VI (text, health coach); Condition VII (text, support coach); Condition VIII (text)
Other: Health Promotion and Education - Digital health tool kit — Receive digital health tool kit
  Other Names: Educational, Digital health tool kit
  Arms: Condition I (text, health kit, health coach, support coach); Condition II (text, health kit, health coach); Condition III (text, health kit, support coach); Condition IV (text, health kit); Condition IX (health kit, health coach, support coach); Condition X (health kit, health coach); Condition XI (health kit, support coach); Condition XII (health kit)
Other: Questionnaires — Quality of Life and Behavioral Questionnaires
  Other Names: Quality of Life Questionnaires

SUMMARY:
This clinical trial studies the effect of four different intervention components "tools" on body weight, nutrition, and physical activity in cancer survivors. Studies indicate that people with a history of cancer whose nutrition and physical activity habits are consistent with the American Cancer Society's Nutrition and Physical Activity Guidelines may have longer disease-free survival. The four different intervention components may help patients with a history of cancer adopt recommended health behaviors after they have completed treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the effect of four candidate intervention components (text messaging, digital health tool kit, health coaching, or support person training), and combinations of the four intervention components, on change cancer survivors' American Cancer Society (ACS) guideline score after 48 weeks of intervention.

SECONDARY OBJECTIVES:

I. To determine the effect of four candidate intervention components (text messaging, digital health tool kit, health coaching, or support person training), and combinations of the four intervention components, on cancer survivors' American Cancer Society (ACS) guideline score after 24 weeks of intervention.

II. To determine the effect of four candidate intervention components, and combinations of the four intervention components, on cancer survivors' intake of fruits and vegetables, whole grains, refined grains, red meat, and processed meats; moderate-to-vigorous physical activity; and body mass index (BMI) after 48 weeks of intervention.

EXPLORATORY OBJECTIVES:

I. To determine the effect of four candidate intervention components (text messaging, digital health tool kit, health coaching, or support person coaching), and combinations of the four intervention components, on cancer survivors' American Cancer Society (ACS) guideline score after 12 weeks of intervention.

II. To describe adherence to each intervention component.

III. To explore the effects of each of the candidate intervention components (text messaging, digital health tool kit, health coaching, support person training) on theoretical constructs (e.g., self-efficacy, outcome expectations, self-monitoring, social support) from 0 to 24 and 48 weeks.

IV. To explore whether sociodemographic (e.g., gender, age, race/ethnicity), clinical (e.g., stage of disease, treatment history, ostomy status, time since diagnosis), and/or psychological/behavioral (e.g., self-efficacy, social support, outcome expectations, depression) factors moderate the intervention components' effects on ACS guideline scores.

VII. To explore change in ACS guideline score in relation to change in fasting insulin, glucose, homeostatic model assessment (HOMA-IR), and inflammatory markers (e.g., Interleukin 6 (IL-6), high-sensitivity C-reactive protein (hs-CRP), Tumor Necrosis Factor alpha (TNF-alpha) for a subset of participants from enrollment to 48 weeks among people with a history of cancer.

VIII. To explore change in ACS guideline score in relation to change in fatigue, depression, and sleep quality from 0 to 24 and 48 weeks among people with a history of cancer.

IX. To explore changes in the ACS guideline score in relation to change in the gut microbiome among a subset of participants with a history of cancer.

X. To describe cancer survivors' 10-year cardiovascular risk using the American Heart Association (AHA) Predicting Risk of cardiovascular disease (CVD) EVENTS (PREVENT) score.

OUTLINE: All patients receive a personal report comparing their nutrition and physical activity to ACS guidelines and a booklet on nutrition and physical activity for patients with a history of cancer. Patients are randomized to 1 of 16 conditions.

CONDITION I: Patients receive text messages and use digital health tool kit for 48 weeks. Patients also receive 13 health coaching sessions over 30 minutes each for 48 weeks. Support persons receive four coaching sessions lasting 30 minutes each, approximately every 12 weeks for 48 weeks.

CONDITION II: Patients receive text messages and use digital health tool kit for 48 weeks. Patients also receive 13 health coaching sessions over 30 each for 48 weeks.

CONDITION III: Patients receive text messages and use digital health tool kit for 48 weeks. Support persons receive four coaching sessions lasting 30 minutes each, approximately every 12 weeks for 48 weeks.

CONDITION IV: Patients receive text messages and use digital health tool kit for 48 weeks.

CONDITION V: Patients receive text messages for 48 weeks. Patients also receive 13 health coaching sessions over 30 minutes each for 48 weeks. Support persons receive four coaching sessions lasting 30 minutes each, approximately every 12 weeks for 48 weeks.

CONDITION VI: Patients receive text messages for 48 weeks. Patients also receive 13 health coaching sessions over 30 minutes each for 48 weeks.

CONDITION VII: Patients receive text messages for 48 weeks. Support persons receive four coaching sessions lasting 30 minutes each, approximately every 12 weeks for 48 weeks.

CONDITION VIII: Patients receive text messages for 48 weeks.

CONDITION IX: Patients use digital health tool kit for 48 weeks. Patients also receive 13 health coaching sessions over 30 minutes each for 48 weeks. Support persons receive four coaching sessions lasting 30 minutes each, approximately every 12 weeks for 48 weeks.

CONDITION X: Patients use digital health tool kit for 48 weeks. Patients also receive 13 health coaching sessions over 30 minutes each for 48 weeks.

CONDITION XI: Patients use digital health tool kit for 48 weeks. Support persons receive four coaching sessions lasting 30 minutes each, approximately every 12 weeks for 48 weeks.

CONDITION XII: Patients use digital health tool kit for 48 weeks.

CONDITION XIII: Patients receive 13 health coaching sessions over 30 minutes each for 48 weeks. Support persons receive four coaching sessions lasting 30 minutes each, approximately every 12 weeks for 48 weeks.

CONDITION XIV: Patients receive 13 health coaching sessions over 30 minutes each for 48 weeks.

CONDITION XV: Support persons receive four coaching sessions lasting 30 minutes each, approximately every 12 weeks for 48 weeks.

CONDITION XVI: Patients receive personal report and booklet only.

ELIGIBILITY:
Inclusion Criteria:

INCLUSION CRITERIA FOR CANCER SURVIVORS:

1. >= 18 years of age.
2. Diagnosis of bladder, breast, colon, endometrial, kidney (renal cell carcinoma), ovarian, prostate, or rectal cancer.
3. Completed all cytotoxic chemotherapy, immunotherapy, targeted therapies, or radiation (if indicated) prior to enrollment. Hormonal treatments are allowed.
4. Owns a smart phone that has access to the Internet and can receive daily text messages.
5. Able to speak and read English or Spanish
6. Have a support person >= 18 years of age who speaks English or Spanish and is willing to provide informed consent and support the participant throughout the study.
7. >= 4 weeks since a major surgery to start of intervention (removal of port or catheter (cath) is not major surgery; reversal of ostomy is major surgery and will require at least 4 weeks prior to enrollment).
8. Readiness, as determined by the Physical Activity Readiness Questionnaire (PAR-Q). If there are any indications that home-based exercise might be unsafe based on PAR-Q, the patient will not be enrolled until confirmation from the patient's provider is received via email and/or phone that they are safe to exercise. Providers do not need to be contacted if patients answer 'yes' to 'Is your doctor currently prescribing any medication for your blood pressure or for a heart condition?

INCLUSION CRITERIA FOR SUPPORT PERSONS:

1. Identified by a cancer survivor participant who has consented to participate in Tools To Be Fit as their support person.
2. 18 years of age or older.
3. Speaks and reads English or Spanish.
4. Consents to complete two online surveys and four 1-on-1 health coaching calls during the 48 week study.

Exclusion Criteria:

EXCLUSION CRITERIA FOR CANCER SURVIVORS:

1. People with potential contraindications to home-based exercise based on the PAR-Q for whom the investigator is unable to obtain physician clearance.
2. ACS guideline score of > 4 out of 6 at enrollment based on self-reported diet, BMI, and physical activity. Our screening survey will ask participants to report their height and weight; usual intake of foods in the ACS guidelines (e.g., red and processed meat, fruits, vegetables, grains); and the Godin Leisure Time Exercise Survey.
3. Used a physical activity tracker and a diet tracking app for >= 1 week in the past 3 months; these are components of our digital health tool kit.
4. Planned major surgery during the study period (removal of port or cath or dermatological procedures excluded)
5. Scheduled to receive any form of cancer therapy during the study period with the exception of hormonal treatments, which are allowed.
6. History of severe cardiovascular, respiratory or musculoskeletal disease or joint problems that preclude moderate physical activity. Examples include unstable angina, recent myocardial infarction, oxygen-dependent pulmonary disease, and osteoarthritis requiring imminent joint replacement. Moderate arthritis that does not preclude physical activity is not a reason for ineligibility.
7. History of psychiatric disorders that would preclude participation in the study intervention (e.g., untreated major depression or psychosis, substance abuse, severe personality disorder) or prevent the patient from giving informed consent.
8. Participating in another weight loss, physical activity or dietary intervention clinical trial. Co-enrollment in some trials involving pharmacologic therapy is allowed. Participants are also allowed to pursue weight loss and physical activity programs on their own, as long as these programs are not provided as part of a clinical trial.
9. Currently pregnant or trying to become pregnant during the study period.
10. Living outside the United States during screening and/or the 48-week study period.

EXCLUSION CRITERIA FOR SUPPORT PERSONS:

1. None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-10-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in American Cancer Society (ACS) guideline score at 48 weeks | Up to 48 weeks
  The ACS Guideline Score is comprised of scores on participant reported food intake (score range from 0-2), physical activity (score range from 0-2), and body mass index (BMI) (score range from 0-2). The total score is calculated by summing the scores on each component with a total score range from 0 to 6. Greater scores indicate a greater level of healthy choices made by the participant. The investigator will assess the independent and interaction effects of the four treatment components on change in ACS score as repeated measures and using a generalized linear mixed effect model, starting with the saturated model, including coefficients for main effects, interactions up to 3-way, and stratification variables (gender and age), and reduce the model via backward variable selection with a 0.05 significance level (alpha(α)=0.05) up to 48 weeks.

SECONDARY OUTCOMES:
Mean change in ACS guideline score at 24 weeks | Up to 24 weeks
  The ACS Guideline Score is comprised of scores on participant reported food intake (score range from 0-2), physical activity (score range from 0-2), and body mass index (BMI) (score range from 0-2). The total score is calculated by summing the scores on each component with a total score range from 0 to 6. Greater scores indicate a greater level of healthy choices made by the participant. The investigator will assess the independent and interaction effects of the four treatment components on change in ACS score as repeated measures and using a generalized linear mixed effect model, starting with the saturated model, including coefficients for main effects, interactions up to 3-way, and stratification variables (gender and age), and reduce the model via backward variable selection with a 0.05 significance level (α=0.05) up to 24 weeks.
Mean change in scores on the individual components of the ACS at 24 weeks | Up to 24 weeks
  The ACS Guideline Score is comprised of individual factor scores on (1) participant reported food intake (score range from 0-2), (2) physical activity (score range from 0-2), and (3) body mass index (BMI) (score range from 0-2). Greater scores indicate a greater level of healthy choices made by the participant. The investigator will assess the independent and interaction effects of the four treatment components on change in the individual ACS guideline factors from 0 to 24 weeks using linear mixed-effects models adjusting for the stratification variables gender and age with the individual factor of interest as the outcome.
Mean change in scores on the individual components of the ACS at 48 weeks | Up to 48 weeks
  The ACS Guideline Score is comprised of individual factor scores on (1) participant reported food intake (score range from 0-2), (2) physical activity (score range from 0-2), and (3) body mass index (BMI) (score range from 0-2). Greater scores indicate a greater level of healthy choices made by the participant. The investigator will assess the independent and interaction effects of the four treatment components on change in the individual ACS guideline factors from 0 to 48 weeks using linear mixed-effects models adjusting for the stratification variables gender and age with the individual factor of interest as the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Van Blarigan, ScD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with research collaborators during the course of the study.
Supporting Information: Study Protocol, SAP

REFERENCES:
- See also: Study Website — https://toolstobefit.eurekaplatform.org/pages/landing?locale=en